CLINICAL TRIAL: NCT06290830
Title: The Effect of Abdominal Massage and Kegel Exercises on Constipation and Quality of Life in Female Students With Functional Constipation: A Randomized Controlled Trial
Brief Title: Abdominal Massage and Kegel Exercises on Constipation and Quality of Life in Female Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sukran Basgol, Assistant Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OMUŞükranBaşgöl01
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Functional Constipation; Constipation; Quality of Life
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Abdominal massage group (Experimental): Abdominal massage is demonstrated by the researchers to a female student with functional constipation. The student will apply exfoliation (superficial and deep), petrissage, and vibration massage movements for about 15 minutes twice a day in the morning and evening hours and at least 30 minutes after the nutritional meal, 5 days a week, for a total of 12 weeks.
  Interventions: Behavioral: Abdominal massage group
- Kegel Exercises group (Experimental): In this group students will perform Kegel exercises; 2 times a day in the morning and evening hours, 5 days a week, for a total of 12 weeks.
  Interventions: Behavioral: Kegel Exercises group
- Both abdominal massage and kegel exercises to gether (Experimental): students will perform both abdominal massage and kegel exercises to gether for a total of 12 weeks
  Interventions: Behavioral: Both abdominal massage and kegel exercises to gether
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Abdominal massage group — abdominal massage creates reflex and mechanical movement of the intestines by applying pressure to the rectum and changing intra-abdominal pressure.
  Arms: Abdominal massage group
Behavioral: Kegel Exercises group — Kegel exercises (also called pelvic floor exercises) have a functional connection with other core muscles and contribute to the synergistic effect of the abdominal and pelvic floor muscles
  Arms: Kegel Exercises group
Behavioral: Both abdominal massage and kegel exercises to gether — with both exercises are performed to accelerate the peristalsis movement by mechanical movements
  Arms: Both abdominal massage and kegel exercises to gether

SUMMARY:
In this prospective, randomized controlled study, n=140 female students with functional constipation studying at two universities Faculty of Health Sciences and meeting the Rome-IV Diagnostic Criteria for Constipation will be included in the study. Between 15.03.2024 and 31.05.2024, n=140 (35=control group, 35=kegel exercise group, 35=abdominal exercise group, 35=abdominal and kegel exercise group) volunteered to participate in the study. Female students with functional constipation will be randomly divided into four groups as intervention and control groups. Personal Information Form", "Bristol Stool Scale", "Constipation Severity Scale", and "Patient Assessment of Constipation Quality of Life Questionnaire" will be used in this study. The scales will be used in the research two times: pre and post-test (scales were reassessed at the end of the study after the exercise intervention). Descriptive statistics, Pearson, and Spearman's correlation analyses will be used in the analysis of research data.

DETAILED DESCRIPTION:
This study aimed to investigate the effect of abdominal massage and kegel exercises on constipation and quality of life in female students with functional constipation.

Type of Research: This study was conducted in a prospective, four-arm, and randomized controlled manner.

Female students with functional constipation studying at two universities Faculty of Health Sciences and meeting the Rome-IV Diagnostic Criteria for Constipation will be included in the study.

The power analysis of this study was performed with G*POWER 3.1.9.7 (Power analysis statistical software). The sample size of the study was based on the average score of the Patient Assessment of Constipation Quality of Life Questionnaire (Patient Assessment of Constipation Quality of Life Questionnaire). It was determined that 31 individuals from each group would be sufficient to participate in the study with an effect size of 0.64, α = 0.05 margin of error, and minimum power = 80% (β = 0.2). Considering the possible missing data, it was calculated that each group should consist of 35 female students with functional constipation with a 10% increase.

Data Collection Tools-Validity and Reliability Information In the study, the "Personal Information Form", "Bristol Stool Scale", "Constipation Severity Scale", and "Patient Assessment of Constipation Quality of Life Questionnaire" will be used. The scales will be used in the research two times: pre and post-test (scales were reassessed at the end of the study after the exercise intervention).

Personal Information Form: The information form developed by the researchers by analyzing the literature consisted of 10 questions about sociodemographic characteristics, health status, and variables affecting constipation.

Bristol Stool Scale: The type of stool is classified into 7 different groups. In the Bristol Stool Scale, the transit time of the stool through the intestine is evaluated over seven different stool types. According to Bristol Stool Scale, 1-2 points are shown as "hard stool", 3-4-5 points as "normal stool" and 6-7 points as "soft-watery stool (diarrhea)".

Constipation Severity Scale: It is a scale for determining the frequency, intensity, and difficulty/difficulty during defecation. In addition, it was aimed to measure the constipation symptoms of the participants through this scale. There are 16 questions on the scale. The scale has three sub-dimensions: fecal obstruction, large bowel laziness, and pain. The score that can be obtained from the Faecal Obstruction sub-dimension is 0-28, the score that can be obtained from the Large Bowel sub-dimension is 0-29, and the score that can be obtained from the Pain sub-dimension is 0-16. The lowest total score that can be obtained from this scale is 0 and the highest score is 73. A high score on the scale indicates that the symptoms are serious. Internal consistency (α = 0.88-0.91) and test-retest reliability (intraclass correlation coefficients = 0.84-0.91) were reported to be high for all subscales.

Patient Assessment of Constipation Quality of Life Questionnaire: This scale measures the quality of life in constipation. This is a 28-item self-assessment scale consisting of "Worry/Anxiety" (11 items), "Physical Discomfort" (4 items), "Psychosocial Discomfort" (8 items), and "Satisfaction" (5 items) subscales. The item scores of the five-point Likert-type scale vary between 1-5. The highest score obtained from the scale is 140 and the lowest score is 28. It is thought that quality of life is negatively affected as the scores obtained from the scale increase. The Cronbach alpha reliability coefficient of the scale is 0.91. The Cronbach alpha reliability coefficient of the "Physical Discomfort" subscale is 0.88, the total item correlation coefficient is 0.91, the Cronbach alpha reliability coefficient of the "Psychosocial Discomfort" subscale is 0.87, the total item correlation coefficient is 0. 82, Cronbach alpha reliability coefficient of "Worry and Anxiety" subscale was 0.85, the total item correlation coefficient was 0.84 and Cronbach alpha reliability coefficient of "Satisfaction" subscale was 0.76, total item correlation coefficient was 0.80.

The female students included in the study will be taught abdominal massage and kegel exercises by the researcher in an appropriate environment according to the interventional group determined as a result of the randomization assignment. The intervention and control groups will be initially trained on nutrition in constipation.

Abdominal massage group (35 students): Abdominal massage is demonstrated by the researchers to a female student with functional constipation. The student will apply exfoliation (superficial and deep), petrissage, and vibration massage movements for about 15 minutes twice a day in the morning and evening hours and at least 30 minutes after the nutritional meal, 5 days a week, for a total of 12 weeks.

Kegel exercise group (35 students): 2 times a day in the morning and evening hours, 5 days a week, for a total of 12 weeks.

Abdominal massage and kegel exercise group (35 students): students will do both abdominal and kegel exercises for 12 weeks

Control group (35 students): No intervention will be made to the control group.

Ethical Aspects of the Research For the ethical suitability of the research, The University Rectorate Ethical approval was obtained at the meeting of the Social and Human Sciences Ethics Committee dated 30.01.2024 and numbered "2023-0844" and written permission was obtained from two universities for data collection. Written informed consent is also obtained from the participating students. The research was conducted following the rules of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

Must include two or more of the following:

* Straining during more than ¼ (25%) of defecations
* Lumpy or hard stools (Bristol Stool Form Scale 1-2) more than ¼ (25%) of defecations
* Sensation of incomplete evacuation of more than ¼ (25%) of defecations
* Sensation of anorectal obstruction/blockage of more than ¼ (25%) of defecations
* Manual maneuvers to facilitate more than ¼ (25%) of defecations (e.g., digital evacuation, support of the pelvic floor)
* Less than 3 defecations per week
* Loose stools are rarely present without the use of laxatives
* Insufficient criteria for irritable bowel syndrome

Exclusion Criteria:

* the study included patients with intra-abdominal infection
* advanced heart disease
* previous bowel surgery
* cancer diagnosis
* irritable bowel syndrome
* any intestinal problem, metabolic, endocrine, and neurological constipation, current or past smoker
* congenital megacolon, pseudo-obstruction, and anorectal disorder
* any mental, psychological, and physical disorder any medication,
* fecal and urinary incontinence,
* pregnant
* do not volunteer to participate in the research will not be included.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Constipation severity change | At baseline and at the end of the day (12 weeks later) of study, constipation severity will assessed.
  As assessed by Constipation Severity Scale, for determining the frequency, intensity, and difficulty/difficulty during defecation. In addition, it was aimed to measure the constipation symptoms of the participants through this scale. There are 16 questions on the scale. The scale has three sub-dimensions: fecal obstruction, large bowel laziness, and pain. The lowest total score that can be obtained from this scale is 0 and the highest score is 73. A high score on the scale indicates that the symptoms are serious.
Quality of Life change | At baseline and at the end of the day (12 weeks later) of study, Quality of Life will assessed.
  As assessed by Patient Assessment of Constipation Quality of Life Questionnaire, for measuring quality of life in constipation. This is a 28-item self-assessment scale consisting of "Worry/Anxiety" (11 items), "Physical Discomfort" (4 items), "Psychosocial Discomfort" (8 items), and "Satisfaction" (5 items) subscales. The highest score that can be obtained from the scale is 140 and the lowest score is 28. It is thought that quality of life is negatively affected as the scores obtained from the scale increase
Bristol stool form score change | At baseline and at the end of the day (12 weeks later) of study, constipation severity will assessed.
  As assessed by Bristol stool form scale is a graded visual scale of stool density from type 1 (hard to pass) to type 7 (the fluid kind). it shows the participant's stool shapes together with precise descriptions regarding form and consistency, and using easily recognizable examples (for example, in type 1, by an illustration of faces as separate balls, a description: "separate hard lumps, like nuts"). In the Bristol Stool Scale, the transit time of the stool through the intestine is evaluated over seven different stool types. According to Bristol Stool Scale, 1-2 points are shown as "hard stool", 3-4-5 points as "normal stool" and 6-7 points as "soft-watery stool (diarrhea)".

IPD SHARING:
Plan to Share IPD: No